CLINICAL TRIAL: NCT07008794
Title: Studying the Effect of Genetic Variation on Efficacy and Safety of Lipid-Lowering Drugs in Patients With Cardiovascular Diseases
Brief Title: Effect of Genetic Variation on Efficacy and Safety of Lipid-Lowering Drugs
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ayad Ali Ahmed Abdullah, PhD candidate in Clinical Pharmacy, Assiut University
Other Study IDs: Statin in cardiovascular
Record Dates: First submitted 2025-05-20; First posted 2025-06-06 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-05

CONDITIONS: Acute Coronary Syndromes
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Atorvastatin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral blood samples (3 mL) were collected in EDTA-containing vacutainer tubes and stored at -80 °C until further analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- The first group=atorvastatin on 40 mg/day,: The first group=atorvastatin on 40 mg/day, the second group = rosuvastatin 20 mg.
  all groups received standard therapy included dual antiplatelets ,ACEIs, beta blockers.
  Interventions: Drug: Atorvastatin 40 mg

INTERVENTIONS:
Drug: Atorvastatin 40 mg — Rosuvastatin 20 mg

SUMMARY:
The primary end point was to reduce LDL-C levels by at least 50%, while the secondary end point was to achieve an LDL-C level below 55 mg/dL. The incidence and specifics of side effects and laboratory abnormalities were recorded throughout the follow-up period to evaluate safeguarding. Liver function tests were performed at baseline and 12 weeks later. Any muscle-related complaints were noted at baseline and during the 12-week sessions. CK total and Hba1c were also assessed

DETAILED DESCRIPTION:
CVD are the world's leading cause of death. Egypt has the largest population among the MENA countries, ranks the 2nd in the region for CVD, accounting for 268.11 deaths, or 32.40% of all deaths. Egypt is also ranked 15th globally for cardiovascular mortality.

The total economic costs from non-communicable illnesses in low- and middle-income countries (LMICs) are anticipated to surpass $7 trillion, representing approximately 4% of their annual output. An estimated $25 billion yearly might be saved by a 10% decrease in mortality from IHD greatly paying the expenses of preventative programs The 2019 and 2023 ESC guidelines state that individuals with ACS should aim for a target LDL-C level of < 55 mg/dL (less than 1.4 mmol/L) and achieve a decrease in LDL-C of at least 50% from the initial level

High-intensity statin regimens are medications that decrease LDL-C concentrations by a minimum of 50% . Some examples of high-intensity regimens include rosuvastatin administered at a dose of 20-40 mg and atorvastatin administered at a dose of 40-80.

Statins have been proven to be safe and well-tolerated in managing ACS. However, high-dose statins occasionally resulted in increased in liver transaminases, particularly ALT, and an elevated frequency of ADR. In addition, the muscular symptoms associated with statin use include clinical rhabdomyolysis and myalgia .

Comparing the effects of high-intensity statins in patients who are globalized after ACS, a topic of numerous investigations recently, rosuvastatin appears to decrease LDL-C levels more effectively than atorvastatin. However, no clinical studies have investigated this issue at Assiut University Heart Hospital. Consequently, this investigation aimed to evaluate the effectiveness and safety of atorvastatin 40 mg and rosuvastatin 20 mg in Egyptian patients who had experienced ACS.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged exceeding 18 years,
* Those with ACS confirmation, and those who had not started statin medication during the last 2 months were included

Exclusion Criteria:

* Patients using bile acid sequestrants (colesevelam, cholestyramine), fenofibrate, ezetimibe, niacin, and/or omega-3, as well as those taking concurrently interacting medications (cyclosporine, gemfibrozil, clarithromycin, and/or itraconazole), were excluded from consideration
* During the recruitment process, the study excluded women who were pregnant, nursing, or of childbearing age without a reliable method of contraception.
* As well as patients with bile duct issues, active liver disease, elevated ALT levels exceeding three times the upper normal limit (UNL), serum creatinine levels above 2 mg/dL,
* Individuals who had undergone or reported a hypersensitivity reaction to any currently used statins

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Initially, the study collected patient information, including smoking status, age, BMI, and sex. Furthermore, concurrent medication use, comorbidities, and a detailed medical history were collected.
  Standard laboratory tests included baseline measurements of HbA1c, blood urea nitrogen, serum creatinine, and whole blood picture. While the following parameters at baseline and after 12 weeks were evaluated: CK, HBA1c, TG, HDL, VLDL-C, and LDL-C. Liver function tests included AST and ALT levels.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
The primary outcome was achieving ≥ 50% LDL-C (mg/dL) reduction from the baseline. | Baseline and 12 weeks
  Group 1; administrate atorvastatin 40 mg while the second group administrated rosuvastatin 20 mg.

SECONDARY OUTCOMES:
Target level | Baseline and 12 weeks
  To achieve attainment of LDL-C level < 55 mg/dL from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Hosam Ali Mohamed, Professor, Study Director — Assiut University
Locations (1):
- Assiut University Heart Hospital, Asyut, Asyut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] WHO. Global causes of deaths. 2021.
- [Background] Byrne RA, Rossello X, Coughlan JJ, Barbato E, Berry C, Chieffo A, Claeys MJ, Dan GA, Dweck MR, Galbraith M, Gilard M, Hinterbuchner L, Jankowska EA, Juni P, Kimura T, Kunadian V, Leosdottir M, Lorusso R, Pedretti RFE, Rigopoulos AG, Rubini Gimenez M, Thiele H, Vranckx P, Wassmann S, Wenger NK, Ibanez B; ESC Scientific Document Group. 2023 ESC Guidelines for the management of acute coronary syndromes. Eur Heart J Acute Cardiovasc Care. 2024 Feb 9;13(1):55-161. doi: 10.1093/ehjacc/zuad107. No abstract available. PMID 37740496
- [Background] Rao SV, O'Donoghue ML, Ruel M, Rab T, Tamis-Holland JE, Alexander JH, Baber U, Baker H, Cohen MG, Cruz-Ruiz M, Davis LL, de Lemos JA, DeWald TA, Elgendy IY, Feldman DN, Goyal A, Isiadinso I, Menon V, Morrow DA, Mukherjee D, Platz E, Promes SB, Sandner S, Sandoval Y, Schunder R, Shah B, Stopyra JP, Talbot AW, Taub PR, Williams MS. 2025 ACC/AHA/ACEP/NAEMSP/SCAI Guideline for the Management of Patients With Acute Coronary Syndromes: A Report of the American College of Cardiology/American Heart Association Joint Committee on Clinical Practice Guidelines. Circulation. 2025 Apr;151(13):e771-e862. doi: 10.1161/CIR.0000000000001309. Epub 2025 Feb 27. PMID 40014670